CLINICAL TRIAL: NCT00876603
Title: A Comparison of Anterior and Posterior Procedures for the Surgical Management of Cervical Spondylotic Myelopathy: Prospective Randomized Clinical Trial
Brief Title: Anterior Vs Posterior Procedures for Cervical Spondylotic Myelopathy: Prospective Randomized Clinical Trial
Acronym: CSM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Professor Keith DK Luk., Department of Orthopaedics and Traumatology, The University of Hong Kong.
Other Study IDs: A Vs P Decompression for CSM
Record Dates: First submitted 2009-04-06; First posted 2009-04-07 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2010-01

CONDITIONS: Cervical Spondylotic Myelopathy
Keywords: cervical spondylotic myelopathy; anterior decompression and fusion; cervical laminoplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- 1
- 2
- CSM - ACDF: Cervical spondylotic myelopathy treated with anterior cervical decompression and fusion
  Interventions: Procedure: ACDF
- CSM - Cervical laminoplasty: Cervical spondylotic myelopathy treated with cervical laminoplasty
  Interventions: Procedure: Cervical laminoplasty

INTERVENTIONS:
Procedure: ACDF — Anterior cervical decompression and fusion
  Groups: CSM - ACDF
Procedure: Cervical laminoplasty — Cervical laminoplasty
  Groups: CSM - Cervical laminoplasty

SUMMARY:
There is no difference in surgical outcomes for patients suffering from cervical spondylotic myelopathy treated with anterior decompression and fusion or posterior cervical laminoplasty.

DETAILED DESCRIPTION:
Cervical spondylotic myelopathy (CSM) is a syndrome consisting of symptoms and signs of cervical spinal cord compression caused by chronic degenerative changes of the cervical spine. CSM is the most serious and disabling condition of cervical spondylosis. Natural history studies showed that most of the CSM patients have a progressive deterioration course and no spontaneous regression occurs. It is suggested that the patients with moderate to severe CSM should be operated as early as possible before neurological deficits are too pronounced.

Although there are many options available for the surgical treatment of cervical spondylotic myelopathy, the choice of surgical approach for CSM is still a controversial issue. Most of the surgeons select the surgical approach based on the number of levels involved and the alignment of the spine. Anterior procedure is generally recommended for patients with compression of less than 3 levels or in patients with kyphotic alignment, while posterior decompression is suggested for three or more levels of compression. Retrospective clinical study however has shown that both anterior and posterior surgeries could produce comparable results. There is no scientific data based on randomized, prospective clinical studies comparing the various surgical alternatives. The existing information does not clearly favor any one single approach or operative option. Since anterior and posterior surgeries carries different risks, it is important to identify the most appropriate surgical procedure that is supported by evidence rather than just by surgeons preference.

The objective of this study is to compare the long-term clinical outcome of anterior approach versus posterior approach in the treatment of cervical myelopathy caused by degenerative disease of the cervical spine.

ELIGIBILITY:
Inclusion Criteria:

* Patients with transverse lesion type of cervical myelopathy caused by cervical spondylosis requiring surgery.
* Involved levels limited to 1, 2 and 3 continuous levels

Exclusion Criteria:

* Radiculomyelopathy
* Cervical kyphosis
* Cervical myelopathy caused by high energy trauma
* Female > 70 years old or patients with severe osteoporosis
* High anaesthetic risk
* Cervical myelopathy other than transverse type
* Cervical myelopathy caused by ossification of posterior longitudinal ligament or inter-vertebral disc herniation.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffer from cervical spondylotic myelopathy requiring surgery.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2001-05; Primary Completion 2010-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Japanese Orthopaedic Association Score for Cervical Myelopathy | 3 months, 6 months, 1 year, 3 years, 5 years and 10 years

SECONDARY OUTCOMES:
Motor and sensory functions, gait and hand functions, neck pain, change in cervical alignment, spinal cord signal change on MRI, operative time, blood loss, duration of in-patient stay, post-operative complication, re-operation rate. | 3 months, 6 months, 1 year, 3 years, 5 years and 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Wai Yuen Cheung, MBBS, FRCS, Principal Investigator — Department of Orthopaedics and Traumatology, The University of Hong Kong; Keith DK Luk, MBBS, FRCS, Study Director — Department of Orthopaedics and Traumatology, The Universityof Hong Kong; Kenneth MC Cheung, MBBS, FRCS, Study Director — Department of Orthopaedics and Traumatology, The University of Hong Kong; Yat Wa Wong, MBBS, FRCS, Principal Investigator — Department of Orthopaedics and Traumatology, The University of Hong Kong.
Locations (1):
- The Duchess of Kent Children's Hospital, Hong Kong, Hong Kong, China